CLINICAL TRIAL: NCT06837051
Title: Protocol for a Randomized Controlled Trial Evaluating the Effect of Modified Olfactory Training on Postoperative Olfactory Dysfunction in Patients With Chronic Rhinosinusitis
Brief Title: The Effect of Modified Olfactory Training on Postoperative Olfactory Dysfunction in Patients With CRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dawei Wu, Associate Researcher, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9059104
Record Dates: First submitted 2025-02-06; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Olfactory Dysfunction; Chronic Rhinosinusitis
Keywords: olfactory dysfunction; chronic rhinosinusitis; endoscopic sinus surgery; olfactory training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Conventional Olfactory Training Group (Active Comparator): Patients are instructed to use the conventional olfactory training device at home twice daily, before breakfast and at bedtime. Four odors will be used: rose, mint, lemon, and clove. In each training session, participants are exposed to each odor for a duration of 10 seconds, followed by a 10-second break before the next odor is presented. Each training session lasts 5 minutes and is conducted for a duration of 12 months. All the patients will be treated with budesonide irrigations. Saline irrigations will be administered twice daily for 12 months using a NeilMed™ (NeilMed, Santa Rosa, CA) squeeze bottle along with salt packets and either distilled or filtered water. 2 mL of 0.5 mg/ 2 mL budesonide (Pulmicort Respules, AstraZeneca Canada, Mis sissauga, ON, Canada) will be added to the irrigation bottles of the patients.
  Interventions: Device: Conventional olfactory training device
- The Modified Olfactory Training Group (Experimental): Patients are instructed to use a modified olfactory training device based on expiratory pressure at home twice daily, before breakfast and at bedtime. Four odors will be used: rose, mint, lemon, and clove. In each training session, participants are exposed to each odor for a duration of 10 seconds, followed by a 10-second break before the next odor is presented. Each training session lasts 5 minutes and is conducted for a duration of 12 months. All the patients will be treated with budesonide irrigations. Saline irrigations will be administered twice daily for 12 months using a NeilMed™ (NeilMed, Santa Rosa, CA) squeeze bottle along with salt packets and either distilled or filtered water. 2 mL of 0.5 mg/ 2 mL budesonide (Pulmicort Respules, AstraZeneca Canada, Mis sissauga, ON, Canada) will be added to the irrigation bottles of the patients.
  Interventions: Device: Modified olfactory training device
- The Control Group (Sham Comparator): Participants will not receive any olfactory training. All the patients will be treated with budesonide irrigations. Saline irrigations will be administered twice daily for 12 months using a NeilMed™ (NeilMed, Santa Rosa, CA) squeeze bottle along with salt packets and either distilled or filtered water. 2 mL of 0.5 mg/ 2 mL budesonide (Pulmicort Respules, AstraZeneca Canada, Mis sissauga, ON, Canada) will be added to the irrigation bottles of the patients.
  Interventions: Drug: Budesonide irrigation

INTERVENTIONS:
Device: Conventional olfactory training device — Four odorants are used: phenyl ethyl alcohol (PEA): rose, menthol: mint, citronellal: lemon, and eugenol: cloves. Training patients will receive four glass vials. Each contains one odorant (5 mL, soaked in cotton pads to prevent spilling) and is labeled with the name of the odorant.
  Budesonide irrigation can effectively target the olfactory cleft area to provide anti-inflammatory effects.
  Arms: The Conventional Olfactory Training Group
Device: Modified olfactory training device — The modified olfactory training device is based on the nasal bidirectional drug delivery system. The device uses breathing pressure to create positive pressure, significantly increasing the deposition rate of odors in the olfactory cleft area.
  Budesonide irrigation can effectively target the olfactory cleft area to provide anti-inflammatory effects.
  Arms: The Modified Olfactory Training Group
Drug: Budesonide irrigation — Budesonide irrigation can effectively target the olfactory cleft area to provide anti-inflammatory effects.
  Arms: The Control Group

SUMMARY:
The goal of this clinical trial is to validate the effectiveness of the modified olfactory training device, the main questions it aims to answer are:

Is it possible that the device can treat postoperative olfactory dysfunction in patients with chronic sinusitis? Compared to the conventional device, how efficient is the modified olfactory training device for treating postoperative olfactory dysfunction in patients with chronic sinusitis?

DETAILED DESCRIPTION:
Endoscopic sinus surgery is an effective treatment for treating olfactory dysfunction related to chronic rhinosinusitis. However, recent studies have shown that most patients experience a return of olfactory function to preoperative levels within months to a year after surgery. Clinically, olfactory training after endoscopic sinus surgery has been proven beneficial for the olfactory recovery.

The improved olfactory training device, based on a nasal bidirectional drug delivery system, can increase the deposition rate in the olfactory fissure region and improve the efficiency of olfactory training.

In this study, the investigators planned to recruit 213 patients and divided them into three groups for control group and olfactory training with conventional and modified devices, and validate the effectiveness of the modified device based on changes in cognitive function and the comparison of the outcomes of the three groups.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of CRSsNP based on the European Position Paper on Rhinosinusitis and Nasal Polyps 2020 (EPOS20).
2. The duration after endoscopic sinus surgery is 3months.
3. Olfactory dysfunction confirmed with the Sniffin's Sticks psychophysical test (TDI score≦30.5) .
4. Willingness to participate in this study and sign the informed consent form (ICF).

Exclusion Criteria:

1. Patients with olfactory impairment due to traumatic, congenital, toxic/drug-induced causes, tumors, or post-upper respiratory infections.
2. Lund-Mackay olfactory cleft score > 0.
3. Patients with severe comorbidities, such as malignant tumors.
4. Current or planned pregnancy prior to the end of study.
5. Patients who are unable to complete the study or are unable to comply with the requirements of the study (such as inability to tolerate olfactory function testing and treatment, memory or behavioral abnormalities, depression, smoking, heavy alcohol use, previous delinquent behavior)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2025-03-14 (Estimated); Primary Completion 2027-03-14 (Estimated); Study Completion 2027-03-14 (Estimated)

PRIMARY OUTCOMES:
The Sniffin's Sticks test | Baseline,Month 3,Month 6,Month 12
  A clinically significant olfactory improvement as measured by Sniffin' Sticks threshold, discrimination, and identification(TDI)( more than 6 scores)

SECONDARY OUTCOMES:
Olfactory cleft CT score | Baseline,Month 3,Month 6,Month 12
Olfactory cleft endoscopy scale (OCES) | Baseline,Month 3,Month 6,Month 12
  The degree of discharge, nasal polyposis, edema, crusting, and scarring scores from 0 to 2 points for each measure. The sum of the olfactory cleft score on both sides is recorded for final results that ranged from 0 to 20 points. Higher scores indicate increased disease severity of the olfactory cleft.
OB volume measurement | Baseline,Month 3,Month 6,Month 12
  MRI scans are performed using a 3T GE scanner with a 8-channel phase-array head coil. OB volumes are obtained by manual bordering and following addition of all slices, which are multiplied by the slice thickness to yield volume.
Questionnaire of Olfactory Disorders - Negative Statements (QOD-NS) | Baseline,Month 3,Month 6,Month 12
  The QOD-NS includes 17 negative statements, each graded from 0 (disagree) to 3 (agree) for a maximum score of 51. Higher QOD-NS scores reflect worse QoL.
Olfactory-Visual Analogue Scale (VAS) | Baseline,Month 3,Month 6,Month 12
  Subjects rate the impact of smell loss on their mood, ability to enjoy food, social interactions, safety, personal hygiene, sex life, ability to cook food, appetite and change in weight from 0 (no impact) to 10 (most impact) for a maximum score of 90. Higher olfactory-VAS scores reflect more severe impacts on daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will decide whether to share the individual participant data after the study.

REFERENCES:
- [Derived] Li Y, Li Y, Zhang Y, Wu D. Protocol for a randomised controlled trial evaluating the effect of modified olfactory training on postoperative olfactory dysfunction in patients with CRS. BMJ Open. 2025 Aug 16;15(8):e101870. doi: 10.1136/bmjopen-2025-101870. PMID 40819876